CLINICAL TRIAL: NCT00766623
Title: Elucidation and Monitoring Postprandial Endothelial Function
Acronym: EMPEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Wageningen universiteit department of human nutrition, Wageningen universiteit
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: NL23651.081.08; empef, abr23651, 08/10 EMPEF
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Cardiovascular Disease; Endothelial Dysfunction
Keywords: endothelium,; postprandial; microvascular; macrovascular
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- High fat meal (Experimental): A high fat milkshake containing 95g of fat
  Interventions: Dietary Supplement: high fat meal
- Control meal (Experimental): Milkshake comparable with a normal breakfast
  Interventions: Dietary Supplement: control meal
- High fat meal 2 (Experimental): A high fat milkshake containing 95g of fat
  Interventions: Dietary Supplement: high fat meal
- High fat meal 3 (Experimental): A high fat milkshake containing 95g of fat
  Interventions: Dietary Supplement: high fat meal
- Control meal 2 (Experimental): Milkshake comparable with a normal breakfast
  Interventions: Dietary Supplement: control meal
- Control meal 3 (Experimental): Milkshake comparable with a normal breakfast
  Interventions: Dietary Supplement: control meal

INTERVENTIONS:
Dietary Supplement: high fat meal — milkshake containing 95g fat
  Arms: High fat meal; High fat meal 2; High fat meal 3
Dietary Supplement: control meal — milkshake comparable with a normal breakfast
  Arms: Control meal; Control meal 2; Control meal 3

SUMMARY:
The primary aim of this study is to evaluate the effect of a high fat challenge on several measures of endothelial function. The secondary aim of this study is to elucidate the mechanism of postprandial endothelial dysfunction and to identify early biomarkers

DETAILED DESCRIPTION:
Endothelial dysfunction (ED) is a hallmark for the initial stage of vascular dysfunction and has been associated with diet-related disorders such as cardiovascular disease. This makes prevention of ED an important health target. From previous studies we know that a high-fat (HF) meal (challenge) impairs postprandial endothelial function (EF). Current studies only evaluated the effect of a HF meal on Flow Mediated Dilatation (FMD), a measure of macro vascular EF. This methodology (FMD) however, is time consuming and large variations in reproducibility are reported in literature. The question remains whether other types of macro- and micro vascular EF measurements can be used to observe ED after a HF meal that are more accurate, faster and easier to perform. In addition, it is know that the postprandial phase results in activation of leukocytes. This activation of leukocytes is likely to contribute to ED, but the exact underling mechanism remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* male, caucasian

Exclusion Criteria: • Allergic to cow milk or dairy products

* Body mass index (BMI) < 18 or > 25 kg/m2
* Urine glucose concentrations outside normal ranges (>0,25 g/l)
* Fasting blood glucose outside the normal range (3 - 5.5 mmol/L)
* Tobacco smoking
* Taking medication or food supplements.
* Received inoculations within 2 months of starting the study or planned to during the study
* Donated or intended to donate blood from 2 months before the study till two months after the study
* Blood Hb values below 8.4 mmol/L
* Diagnosed with any long-term medical condition (e.g., diabetes, hemophilia, cardiovascular disease, anemia, gastrointestinal disease, renal failure)
* High blood pressure (systolic BP> 140 mmHg and/or diastolic BP>90 mmHg)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Macrovascular local arterial stiffness by echo-tracking | 0, 3, 6 hours
Macrovascular regional arterial stiffness by tonometry | 0, 3, 6 h
Macrovascular circulation by flow mediated dilatation | 0, 3, 6h
Microvascular circulation by iontophoresis/laser doppler | 0, 3, 6h

SECONDARY OUTCOMES:
PBMC gene expression profiles | 0, 1, 2, 3, 5, 6 hours
Leukocyte activation markers | 0, 3, 6h
cytokine profiles | 0, 1, 2, 3, 5, 6 hours
known plasma markers of ED | 0, 1, 2, 3, 5, 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Müller, Prof.Dr, Study Chair — Chair Department of human nutrition NMG group; Lydia A Afman, PhD, Study Director — Senior scientist department Human Nutrition Wageningen University
Locations (1):
- Wageningen universiteit division of human, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] Esser D, Oosterink E, op 't Roodt J, Henry RM, Stehouwer CD, Muller M, Afman LA. Vascular and inflammatory high fat meal responses in young healthy men; a discriminative role of IL-8 observed in a randomized trial. PLoS One. 2013;8(2):e53474. doi: 10.1371/journal.pone.0053474. Epub 2013 Feb 6. PMID 23405070